CLINICAL TRIAL: NCT06057948
Title: Phase II Trial of a Bivalent Vaccine With the Immunological Adjuvant OPT-821 (QS-21), in Combination With Randomization of Oral β-glucan, for High-Risk Neuroblastoma
Brief Title: A Study of a Vaccine in Combination With Beta-glucan in People With Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-198
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Neuroblastoma; High-risk Neuroblastoma; Metastatic Neuroblastoma
Keywords: Neuroblastoma; High-risk Neuroblastoma; Metastatic Neuroblastoma; HR-NB; Memorial Sloan Kettering Cancer Center; 23-198
MeSH Terms: conditions — Neuroblastoma | interventions — saponin QA-21V1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will receive oral β-glucan (40 mg/kg/day) for 14 days on, and 14 days off, beginning with vaccination #1 and continuing until vaccination #5 (~20 weeks), then only one 14-day cycle with each of vaccinations #6-#10.
  Interventions: Biological: OPT-821 (QS-21); Dietary Supplement: oral β-glucan
- Group 2 (Experimental): Participants will receive oral β-glucan (40 mg/kg/day) for 14 days on, and 14 days off, beginning with vaccination #1 and continuing until vaccination #7 (~52 weeks), then only one 14-day cycle with each of vaccinations #8-#10.
  Interventions: Biological: OPT-821 (QS-21); Dietary Supplement: oral β-glucan

INTERVENTIONS:
Biological: OPT-821 (QS-21) — Comprised of the immunological adjuvant OPT-821 (QS-21)
Dietary Supplement: oral β-glucan — Participants will be randomized to receive this agent in two different schedules

SUMMARY:
The purpose of this study is to test which treatment schedule of β-glucan with bivalent vaccine is more effective for participants with high-risk neuroblastoma that is in complete remission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by international criteria,102 i.e., histopathology (confirmed by the MSK Department of Pathology) or BM metastases plus high urine catecholamine levels, or positivity in MIBG scan.
* HR-NB as defined by risk-related treatment guidelines and international criteria,102 i.e., metastatic/non-localized disease with MYCN amplification (any age), metastatic disease >18 months old, MYCN-amplified localized disease (any age), or disease resistant to standard chemotherapy.
* HR-NB (as defined above) and in 1) first CR at ≥ 6 months from initiation of immunotherapy using anti-GD2 antibody, or 2) second or subsequent CR (achieved after treatment for PD). CR is defined according to the International Neuroblastoma Response Criteria. Patients with positive MIBG scan but negative FDG-PET scan, and CR in BM, are eligible.
* Patients with grade 3 toxicities or less using the Common Toxicity Criteria (Version 5.0) developed by the National Cancer Institute of the USA (CTCAE v5.0) related to hematologic, cardiac, neurological, pulmonary, renal, hepatic or gastrointestinal function as determined by blood tests or physical exam. Plus:

  * Absolute neutrophil count (ANC) ≥ 500/mcl
  * Absolute lymphocyte count ≥ 500/mcl
* >21 and <180 days between completion of systemic therapy and 1st vaccination.
* A negative pregnancy test is required for patients with child-bearing capability
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Patients with grade 4 hematologic, cardiac, neurological, pulmonary, renal, hepatic or gastrointestinal function as determined by blood tests or physical exam, using the Common Toxicity Criteria (Version 5.0) developed by the National Cancer Institute of the USA.
* History of allergy to KLH, QS-21, OPT-821, or glucan
* Prior treatment with this vaccine.
* Active life-threatening infection requiring systemic therapy.
* Inability to comply with protocol requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Mean antibody titer in ng/ml of anti-GD2 IgG1 titer | up to 32 weeks
  To determine the effect of oral β-glucan schedule on anti-GD2 antibody titers among patients who are in first or second (or later) CR, i.e., have no evidence of neuroblastoma by standard studies.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org